CLINICAL TRIAL: NCT04760418
Title: Evaluating the Impact of Trauma, Trauma-Focused Therapy Services, and COVID-19 Among Patients in the University of Kentucky SMART Clinic
Brief Title: Trauma and Trauma-Focused Therapy in the University of Kentucky SMART Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christal L Badour (Other)
Responsible Party: Sponsor-Investigator, Christal L Badour, Assistant Professor of Psychology, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 64485
Record Dates: First submitted 2021-02-10; First posted 2021-02-18 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: PTSD; Opioid-use Disorder; Substance Use Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Non-Concurrent Multiple Baseline Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4 week baseline (Experimental): Participants in this arm are randomized to a 4-week baseline period with repeated weekly assessment after the initial intake. This is followed by 12 sessions of weekly individual manualized Concurrent Treatment of PTSD and Substance Use Disorders Using Prolonged Exposure (COPE)
  Interventions: Behavioral: Concurrent Treatment of PTSD and Substance Use Disorders Using Prolonged Exposure (COPE)
- 6 week baseline (Experimental): Participants in this arm are randomized to a 6-week baseline period with repeated weekly assessment after the initial intake. This is followed by 12 sessions of weekly individual manualized Concurrent Treatment of PTSD and Substance Use Disorders Using Prolonged Exposure (COPE)
  Interventions: Behavioral: Concurrent Treatment of PTSD and Substance Use Disorders Using Prolonged Exposure (COPE)

INTERVENTIONS:
Behavioral: Concurrent Treatment of PTSD and Substance Use Disorders Using Prolonged Exposure (COPE) — A 12-session integrated cognitive behavioral therapy for posttraumatic stress disorder and substance use

SUMMARY:
Opioid misuse is a national public health epidemic. More than 130 people in the United States die each day following an opioid overdose, and over 2 million people meet criteria for an opioid use disorder (OUD). Medication-assisted treatment (MAT), which involves use of medication (buprenorphine, methadone, naltrexone) in combination with behavioral therapy or counseling, is the most effective intervention for OUD. Yet, MAT remains less than optimally effective, particularly for patients with psychiatric comorbidity [6]. Novel approaches are needed to improve long-term outcomes for OUD patients.

Psychological trauma and posttraumatic stress disorder (PTSD) are highly prevalent among individuals with OUD. Over 90% of adults with OUD report a lifetime history of trauma. Among OUD patients engaged in MAT, nearly 20% report experiencing at least one new traumatic event each month, and nearly a third meet criteria for a co-occurring diagnosis of posttraumatic stress disorder (PTSD). Several studies have linked new incidents of trauma as well as the presence of PTSD to poorer MAT engagement and poorer treatment outcomes, including treatment interruption and premature dropout. Preliminary evidence suggests that engaging in trauma-focused treatment for PTSD concurrent with MAT may result in better long-term adherence to medication for OUD. However, recent evidence finds that fewer than half of patients with PTSD in MAT receive any trauma-focused treatment, and even fewer receive evidence-based interventions.

Trauma-focused treatments that concurrently address symptoms of PTSD and substance abuse using an integrated approach have been recommended over traditional substance abuse interventions for patients with this complex dual diagnosis presentation. Concurrent Treatment of PTSD and Substance Use Disorders Using Prolonged Exposure (COPE) is a 12-session evidence-based cognitive-behavioral therapy that integrates exposure therapy for PTSD with cognitive-behavioral skills for addressing problem substance use. COPE has demonstrated efficacy for reducing symptoms of PTSD and substance use disorder across multiple trials. Most samples have included patients with alcohol use disorder or mixed substance use disorder diagnoses. The proposed pilot study would collect preliminary feasibility data to support the first trial of COPE for patients with OUD (and other substance use disorders) who are currently engaged in MAT. As such, a primary aim of the current pilot is to obtain patient feedback regarding the acceptability and applicability of COPE for patients with PTSD receiving MAT treatment through the Supportive Medication Assisted Recovery Treatment (SMART) Program within the University of Kentucky (UK) Department of Psychiatry, an outpatient buprenorphine clinic. The investigators believe that it is critical to engage patients directly in the process of intervention development/refinement to determine how an existing evidence-based intervention like COPE might be modified to best fit the unique needs of patients receiving MAT.

DETAILED DESCRIPTION:
All patients served by the SMART clinic in UK Psychiatry will be invited to complete an online survey to assess for lifetime history of trauma, current PTSD symptoms perceptions of how patients' trauma history and PTSD symptoms are related to their substance use (e.g., do they perceive there to be a connection) and other mental health problems, whether patients have received treatment directly focused on trauma and/or PTSD symptoms and if so how helpful they perceived this treatment to be, and patient interest in receiving additional individual trauma-focused treatment as part of their care within the SMART program.

Patients indicating interest in trauma-focused treatment will be provided with additional details regarding the purpose of the pilot trial to obtain patient feedback regarding their impressions of the 12-session COPE intervention, and feedback regarding how the treatment could be modified to better meet the needs of patients in the UK Psychiatry SMART Program and other MAT programs. Information regarding patient recovery is collected and retained within an internal database within the SMART program to track patient recovery services week-to-week as part of routine clinical services. This database is retained on secured computer systems within the clinic. The investigators will seek permission from participants to draw the following historical information from this database and link it to the survey responses they provide as part of this research study to allow us to examine whether the following clinical factors differ as a function of trauma history or PTSD symptoms:

* Dates of scheduled and attended visits (length and frequency of care)
* Results of urine drug screens
* Weekly report of substance use, mental health, physical pain, and recovery activities (See attached Recovery Update Form)
* Medications patients are taking
* Emergency department visits or hospitalizations since beginning treatment In addition, patients with probable PTSD on the PCL-5 who express interest in participating in the pilot trial will be invited to complete clinical interviews at baseline to assess for PTSD diagnosis/severity and co-occurring conditions that would contraindicate participation in the treatment portion of the study (i.e., schizophrenia or other psychotic disorders, current manic episode, acute suicidal ideation with intent). A total of 6 patients with a current diagnosis of PTSD (who are deemed not at high risk for suicide, have been actively engaged in MAT for at least 4 weeks, and are determined to be medically stable) will be invited to participate in the pilot trial. Eligible patients will then complete additional baseline interviews to assess substance use frequency/quantity, SUD and depression diagnoses, and qualitative information regarding participants' beliefs regarding the role of trauma and PTSD symptoms in their recovery, satisfaction with prior treatment experience, and expectations regarding their experience with COPE.

The treatment part of the study will utilize a randomized, non-concurrent multiple baseline design across participants. This is a form of single-case experimental design that provides a time and cost-effective method of evaluating initial efficacy or effectiveness of an intervention while controlling for the passage of time and repeated assessment in small numbers of patients. Patients will be randomized to either a 4- (n=3) or 6-week (n =3) baseline assessment phase where weekly self-report measures of PTSD symptoms will be completed prior to initiating the COPE treatment. Randomizing to varying baseline periods enables assessments of whether symptoms change (only or more rapidly) when the COPE intervention is applied (i.e., each participant acts as their own control). This design allows for causal inferences and controls for many threats to internal validity. Dr. Badour (PI) will train and supervise clinical psychology doctoral student therapists in delivery of the COPE intervention. Patients will meet with an independent assessor at three points throughout the treatment (3 visits at baseline, 1 visit after session 6, and 2 visits after session 12) to assess symptoms and to provide both quantitative and qualitative feedback regarding their preferences and perspective on the treatment (e.g., treatment credibility, clarity and applicability of material, patient satisfaction, therapeutic alliance) and ways the content could be modified to better fit their needs. At the session 12 assessment, interview measures of PTSD and depression symptoms will be repeated to assess symptom change. Self-report symptoms of PTSD and depression will be administered weekly throughout treatment. MAT adherence and substance use will be monitored as part of routine clinical procedures in the SMART program using the attached Recovery Update Form. As not all patients are seen weekly at the SMART Program, the Recovery Update Form will be administered by the research team on weeks when patients do not have regular clinic visits. The addition of up to two "stressor" sessions (for 14 total possible sessions) will be offered. Content of these sessions will be allowed to deviate from the protocol to address current stressors that arise during the course of treatment. A previous psychotherapy trial found that this modification increases flexibility in PTSD treatment without sacrificing efficacy, and is more in line with a patient-centered approach to treatment. With the exception of the addition of COPE, MAT and other therapeutic programming will continue per normal (e.g., group medication management, ongoing therapy groups, case management). Clinical and demographic data collected by providers in the course of treatment will be obtained and examined for its relevance to illness course and treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Currently a patient in the University of Kentucky Department of Psychiatry Supportive Medication and Recovery Treatment (SMART) Program for at least 4 weeks
* Current diagnosis PTSD

Exclusion Criteria:

* History of schizophrenia or other psychotic disorder
* Current mania

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | Average symptom level and change slope from start to end of baseline (4 or 6 weeks) vs. from start to end of the 12-week treatment period
  Change in Posttraumatic Stress Disorder Symptom Severity
Recovery Update Form | Average symptom level and change slope from start to end of baseline (4 or 6 weeks) vs. from start to end of the 12-week treatment period
  Frequency of Substance Use

CONTACTS AND LOCATIONS:
Overall Officials: Christal Badour, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication and are de-identified will be shared with investigators upon request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be shared upon request from investigators beginning immediately after publication
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] CDC, National Vital Statistics System, Mortality. CDC WONDER, Atlanta, GA: US Department of Health and Human Services. https://wonder.cdc.gov. 2018.
- [Background] Hughes, A., et al., Prescription drug use and misuse in the United States: Results from the 2015 National Survey on Drug Use and Health. NSDUH Data Review, A1-A24. 2016.
- [Background] Rudd RA, Seth P, David F, Scholl L. Increases in Drug and Opioid-Involved Overdose Deaths - United States, 2010-2015. MMWR Morb Mortal Wkly Rep. 2016 Dec 30;65(50-51):1445-1452. doi: 10.15585/mmwr.mm655051e1. PMID 28033313
- [Background] SAMHSA, 2016 National Survey on Drug Use and Health. . 2016.
- [Background] Oesterle TS, Thusius NJ, Rummans TA, Gold MS. Medication-Assisted Treatment for Opioid-Use Disorder. Mayo Clin Proc. 2019 Oct;94(10):2072-2086. doi: 10.1016/j.mayocp.2019.03.029. Epub 2019 Sep 19. PMID 31543255
- [Background] National Academies of Sciences, Engineering, and Medicine; Health and Medicine Division; Board on Health Sciences Policy. Medication-Assisted Treatment for Opioid Use Disorder: Proceedings of a Workshop-in Brief. Washington (DC): National Academies Press (US); 2018 Nov 30. Available from http://www.ncbi.nlm.nih.gov/books/NBK534504/ PMID 30507113
- [Background] Lawson KM, Back SE, Hartwell KJ, Moran-Santa Maria M, Brady KT. A comparison of trauma profiles among individuals with prescription opioid, nicotine, or cocaine dependence. Am J Addict. 2013 Mar-Apr;22(2):127-31. doi: 10.1111/j.1521-0391.2013.00319.x. PMID 23414497
- [Background] Peirce JM, Brooner RK, King VL, Kidorf MS. Effect of traumatic event reexposure and PTSD on substance use disorder treatment response. Drug Alcohol Depend. 2016 Jan 1;158:126-31. doi: 10.1016/j.drugalcdep.2015.11.006. Epub 2015 Nov 21. PMID 26652898
- [Background] Ecker AH, Hundt N. Posttraumatic stress disorder in opioid agonist therapy: A review. Psychol Trauma. 2018 Nov;10(6):636-642. doi: 10.1037/tra0000312. Epub 2017 Jul 31. PMID 28758767
- [Background] Hien DA, Nunes E, Levin FR, Fraser D. Posttraumatic stress disorder and short-term outcome in early methadone treatment. J Subst Abuse Treat. 2000 Jul;19(1):31-7. doi: 10.1016/s0740-5472(99)00088-4. PMID 10867298
- [Background] Meshberg-Cohen S, Black AC, DeViva JC, Petrakis IL, Rosen MI. Trauma treatment for veterans in buprenorphine maintenance treatment for opioid use disorder. Addict Behav. 2019 Feb;89:29-34. doi: 10.1016/j.addbeh.2018.09.010. Epub 2018 Sep 12. PMID 30243036
- [Background] Moreland, A., K. Crum, and C. Newman, Comorbid PTSD among women with opioid use disorder: Prevalence of symptoms and utilization in trauma-focused treatment, in International Society for Traumatic Stress Studies annual meeting. 2019: Boston, MA.
- [Background] Roberts NP, Roberts PA, Jones N, Bisson JI. Psychological interventions for post-traumatic stress disorder and comorbid substance use disorder: A systematic review and meta-analysis. Clin Psychol Rev. 2015 Jun;38:25-38. doi: 10.1016/j.cpr.2015.02.007. Epub 2015 Mar 3. PMID 25792193
- [Background] Simpson TL, Lehavot K, Petrakis IL. No Wrong Doors: Findings from a Critical Review of Behavioral Randomized Clinical Trials for Individuals with Co-Occurring Alcohol/Drug Problems and Posttraumatic Stress Disorder. Alcohol Clin Exp Res. 2017 Apr;41(4):681-702. doi: 10.1111/acer.13325. Epub 2017 Feb 10. PMID 28055143
- [Background] Back SE, Killeen T, Badour CL, Flanagan JC, Allan NP, Ana ES, Lozano B, Korte KJ, Foa EB, Brady KT. Concurrent treatment of substance use disorders and PTSD using prolonged exposure: A randomized clinical trial in military veterans. Addict Behav. 2019 Mar;90:369-377. doi: 10.1016/j.addbeh.2018.11.032. Epub 2018 Nov 27. PMID 30529244
- [Background] Brady KT, Dansky BS, Back SE, Foa EB, Carroll KM. Exposure therapy in the treatment of PTSD among cocaine-dependent individuals: preliminary findings. J Subst Abuse Treat. 2001 Jul;21(1):47-54. doi: 10.1016/s0740-5472(01)00182-9. PMID 11516926
- [Background] Mills KL, Teesson M, Back SE, Brady KT, Baker AL, Hopwood S, Sannibale C, Barrett EL, Merz S, Rosenfeld J, Ewer PL. Integrated exposure-based therapy for co-occurring posttraumatic stress disorder and substance dependence: a randomized controlled trial. JAMA. 2012 Aug 15;308(7):690-9. doi: 10.1001/jama.2012.9071. PMID 22893166
- [Background] Norman SB, Trim R, Haller M, Davis BC, Myers US, Colvonen PJ, Blanes E, Lyons R, Siegel EY, Angkaw AC, Norman GJ, Mayes T. Efficacy of Integrated Exposure Therapy vs Integrated Coping Skills Therapy for Comorbid Posttraumatic Stress Disorder and Alcohol Use Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2019 Aug 1;76(8):791-799. doi: 10.1001/jamapsychiatry.2019.0638. PMID 31017639
- [Background] Persson A, Back SE, Killeen TK, Brady KT, Schwandt ML, Heilig M, Magnusson A. Concurrent Treatment of PTSD and Substance Use Disorders Using Prolonged Exposure (COPE): A Pilot Study in Alcohol-dependent Women. J Addict Med. 2017 Mar/Apr;11(2):119-125. doi: 10.1097/ADM.0000000000000286. PMID 28079572
- [Background] Ruglass LM, Lopez-Castro T, Papini S, Killeen T, Back SE, Hien DA. Concurrent Treatment with Prolonged Exposure for Co-Occurring Full or Subthreshold Posttraumatic Stress Disorder and Substance Use Disorders: A Randomized Clinical Trial. Psychother Psychosom. 2017;86(3):150-161. doi: 10.1159/000462977. Epub 2017 May 11. PMID 28490022